CLINICAL TRIAL: NCT04561622
Title: Emotional Proactive Processing in Bipolar Disorder
Acronym: PROEMO_BP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.387; 2019-A03026-51 (Other: ID RCB)
Record Dates: First submitted 2020-08-12; First posted 2020-09-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Disorder; Bipolar I Disorder; Bipolar II Disorder
Keywords: bipolar disorder; emotion; cognition; stroop; proactive emotional processing
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bipolar patients: Bipolar patients (type I,II, NOS) of the bipolar disorder expert center of CHU Grenoble Alpes.
  Interventions: Behavioral: Emotional Stroop Task
- Healthy controls: Volunteers without any psychiatric disease matching inclusion criteria
  Interventions: Behavioral: Emotional Stroop Task

INTERVENTIONS:
Behavioral: Emotional Stroop Task — Classic Stroop task The subject names one of the 3 colors of the crosses on a sheet.Then, the subject must read the words written on the sheet for 45 seconds.These are the words: RED, BLUE and GREEN, written in black color. The subject must name the color of the word.
  Emotional Stroop task This is a computed task in which the patient is asked to answer both as accurately and as quickly as possible.
  The target stimulus is an emotional face of joy or anger, surmounted by the word "joy" or "anger".The subject must respond using the arrow corresponding to the face he sees.
  A training phase is offered to the subject.
  3 / Categorization task For each trial the participant will visualize a short emotional film or not. Then, the participant will have to choose, the emotion corresponding to what he just saw. A training period is offered too.
  Other Names: Classic Stroop Task; Categorization of Emotional Stimuli Task

SUMMARY:
The main objective of this project is to identify behavioral specificities of the proactive emotional brain among bipolar patients, compared to healthy subjects. These could contribute to some of the emotional processing biases that can be observed in these patients. To achieve this goal, two behavioral tasks will be administer (emotional stroop and emotional stimuli categorization task) to bipolar patients and control subjects, and their performances will be compared.

DETAILED DESCRIPTION:
This is a case-control non-interventional study comparing bipolar patients to matched healthy controls during one assessment visit at the University Hospital of Grenoble.

The experimentation phase takes place in three stages: first, the experimenter collects demographic data (age and level of study, lack of medical history and treatments that may interfere with the task). For bipolar subjects, it also collects the type of bipolarity, the type and date of the last episode, the age of the onset of the disease and the treatment.

Secondly, the subject performs a classic Stroop task lasting 3 to 5 minutes, including instructions.

Finally, the subject performs the two main tasks: the emotional Stroop task lasting about 20 minutes and then the task of emotional stimuli categorization lasting about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Francophones
* Bipolar disorder diagnosis (for patients) according to DSM-5 / CIM-10 criteria
* Affiliation to the French social security insurance

Exclusion Criteria:

* uncorrected perceptual disturbance
* psychiatric disorders other than bipolarity as the main psychiatric disorder or a condition which may affect the tasks proposed for the patients' group
* subject under legal protection
* subject deprived of freedoms by a judicial or administrative decision
* drug abuse less than 12 hours before the assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: bipolar patients cohort followed-up in the Expert Center of University Hospital of Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
performances at the emotional Stroop task | day1
  percentage of correct answers ( in %), reaction time ( in seconds) and inverse efficiency score ( N.A)

SECONDARY OUTCOMES:
sensitivity to interference during Stroop tasks | day1
  -reaction time (in seconds) in the different conditions of the task (reading in the congruent condition, interference during the incongruent condition)
Effect of mood state (depressive state) on behavioral tasks' performances | day 1
  assessment of the impact of mood scales (MADRS) scores on behavioral tasks performances
Effect of mood state (hypo/manic state) on behavioral tasks' performances | day 1
  assessment of the impact of mood scales (YMRS) scores on behavioral tasks performances

CONTACTS AND LOCATIONS:
Overall Officials: Mircea Polosan, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, La Tronche, Isère, France

IPD SHARING:
Plan to Share IPD: Undecided
If the patient accepts all the characteristics useful for the study will be available in our results.

REFERENCES:
- [Background] Beffara B, Wicker B, Vermeulen N, Ouellet M, Bret A, Molina MJ, Mermillod M. Reduction of interference effect by low spatial frequency information priming in an emotional Stroop task. J Vis. 2015;15(6):16. doi: 10.1167/15.6.16. PMID 26024463
- [Background] Golden, C. (1978). Diagnosis and Rehabilitation in Clinical Neuropsychology. College of Psychology: Faculty Books and Book Chapters. https://nsuworks.nova.edu/cps_facbooks/48